CLINICAL TRIAL: NCT00978692
Title: Toric Orthokeratology for Slowing Eye Elongation in Astigmatic Children
Brief Title: Toric Orthokeratology - Slowing Eye Elongation
Acronym: TO-SEE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Collaborators: Menicon Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Pauline Cho, Professor, The Hong Kong Polytechnic University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H-ZG30
Record Dates: First submitted 2009-09-16; First posted 2009-09-17 (Estimated); Last update posted 2016-02-22 (Estimated); Status verified 2016-02

CONDITIONS: Myopia; Astigmatism
Keywords: Myopia; Astigmatism; Orthokeratology; Corneal thickness; Corneal curvatures; Corneal biomechanics
MeSH Terms: conditions — Myopia; Astigmatism | interventions — Eyeglasses

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Toric orthokeratology lenses (Experimental): Children wearing toric ortho-k lenses at night for correcting astigmatism and myopia will be the study group
  Interventions: Device: Toric Orthokeratology lenses
- Single-vision spectacles (Other): Children wearing single-vision spectacles in the daytime for correcting the refractive error will be serve as control group
  Interventions: Device: Single-vision spectacles

INTERVENTIONS:
Device: Toric Orthokeratology lenses — Children wearing toric orthokeratology at night for correcting astigmatism and myopia will be the study group
  Other Names: corneal reshaping therapy
  Arms: Toric orthokeratology lenses
Device: Single-vision spectacles — Children wearing single-vision spectacles in the daytime for correcting the refractive errors will serve as the control group
  Other Names: glasses
  Arms: Single-vision spectacles

SUMMARY:
The aims of this study are to investigate the effects of ortho-k for astigmatic and myopic reduction and myopic control in children, and the long term effects on corneal curvatures and biomechanics.

DETAILED DESCRIPTION:
Ortho-k has been shown to be effective in correcting low myopia but relatively ineffective for astigmatism, using spherical reverse geometry lens designs. Toric ortho-k lenses have been introduced in recent years but the efficacy for astigmatic reduction and for myopic control in children have not been confirmed. The mechanism of myopic reduction in ortho-k cannot be fully explained by changes to the anterior corneal curvatures. It is therefore possible that other corneal parameters such as posterior corneal curvature and corneal biomechanics may contribute to the mechanism.

The current study aims at investigating the efficacy of toric ortho-k lenses for correcting myopic astigmatism and for retarding myopic progression in children compared to children wearing single-vision spectacles. Long term changes to other corneal parameters such as posterior cornea curvatures, topographical corneal thickness, corneal hysteresis, corneal resistance factor, with and without ortho-k lens wear will also be investigated.

ELIGIBILITY:
Inclusion Criteria:

* Myopia (refractive sphere): more than -0.50DS to -5.00DS
* Astigmatism: with-the-rule astigmatism more than -1.25DC
* Anisometropia: ≤ 1.50D in both refractive sphere
* Best corrected monocular visual acuity: equal to or better than 0.10 in logMAR scale in both eyes
* Availability for follow-up for at least 2 years

Exclusion Criteria:

* Strabismus at distance or near
* Contraindication for contact lens wear and orthokeratology (e.g. limbus to limbus corneal cylinder and dislocated corneal apex
* Prior experience with the use of rigid lenses (including orthokeratology)
* Prior experience with myopia control treatment (e.g. refractive therapy or progressive spectacles)
* Systemic or ocular conditions which may affect contact lens wear (e.g. allergy and medication)
* Systemic or ocular conditions which may affect refractive development (e.g. Down syndrome, ptosis)

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 80 (Actual)
Dates: Start 2008-05; Primary Completion 2012-07 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
To determine the eyeball elongation in children wearing ortho-k lenses | Before lens wear, 6, 12,18, 24 months after lens wear

SECONDARY OUTCOMES:
To determine the posterior corneal curvatures, topographic corneal thickness, corneal volume, corneal hysteresis and corneal resistance factor in a group of children and compare these parameters with the ortho-k children | Before lens wear, 6, 12,18, 24 months after lens wear
To investigative the efficacy of toric orthokeratology for correcting astigmatism and myopia | Before lens wear, 6, 12,18, 24 months after lens wear

CONTACTS AND LOCATIONS:
Overall Officials: Pauline Cho, PhD, Principal Investigator — The Hong Kong Polytechnic University
Locations (1):
- School of Optometry, The Hong KOng Polytechnic University, Hong Kong SAR, China

REFERENCES:
- [Background] Chen C, Cheung SW, Cho P. Myopia control using toric orthokeratology (TO-SEE study). Invest Ophthalmol Vis Sci. 2013 Oct 3;54(10):6510-7. doi: 10.1167/iovs.13-12527. PMID 24003088
- [Background] Chen CC, Cheung SW, Cho P. Toric orthokeratology for highly astigmatic children. Optom Vis Sci. 2012 Jun;89(6):849-55. doi: 10.1097/OPX.0b013e318257c20f. PMID 22561203
- [Background] Chen C, Cho P. Toric orthokeratology for high myopic and astigmatic subjects for myopic control. Clin Exp Optom. 2012 Jan;95(1):103-8. doi: 10.1111/j.1444-0938.2011.00616.x. Epub 2011 Sep 5. No abstract available. PMID 21895768